CLINICAL TRIAL: NCT06741722
Title: Safety and Efficacy of Mitoxantrone Hydrochloride Liposome Based DCMG Regimen for Relapsed/refractory Acute Myeloid Leukemia
Brief Title: Safety and Efficacy of Mitoxantrone Hydrochloride Liposome Based DCMG Regimen for R/R AML
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Ning Gao, Chief Physician, Beijing 302 Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AML_DCMG_2024
Record Dates: First submitted 2024-12-09; First posted 2024-12-19 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: AML; Relapsed Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
Keywords: AML; mitoxantrone liposome; Acute Myeloid Leukemia; relapsed/refractory AML; DCMG chemotherapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine; Azacitidine; Cytarabine; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DCMG (Experimental): Patients are treated with DCMG chemotherapy regimen.
  Interventions: Drug: Decitabine, Azacitidine, Mitoxantrone liposome, Cytarabine, G-CSF

INTERVENTIONS:
Drug: Decitabine, Azacitidine, Mitoxantrone liposome, Cytarabine, G-CSF — The specific administration times and dosages for the DCMG chemotherapy regimen are as follows:
  M: Mitoxantrone Hydrochloride Liposome Injection: 15 mg/m², IV, on Day 1, every 4 weeks (q4w); D: Decitabine: 20 mg/m², IV, Days 1-5, q4w; (or Azacitidine: 75 mg/m², IV, Days 1-7, q4w); C: Cytarabine: 100 mg, IV, every 12 hours on Days 1-5, q4w; For patients with hypoplastic bone marrow, the dose of cytarabine injection is 10 mg, every 12 hours, q4w; G: G-CSF: 5 μg/kg, subcutaneous injection, from Day 0 until the white blood cell count exceeds 10.0×10^9/L, at which point chemotherapy is stopped; or Pegylated Recombinant Human Granulocyte Stimulating Factor Injection: 100 μg/kg, subcutaneous injection, on Day 0.
  One cycle lasts for 4 weeks, with a planned administration of 1 or 2 cycles.

SUMMARY:
The DCMG regimen includes decitabine or azacitidine (hypomethylating agents), mitoxantrone liposome, cytarabine, and granulocyte colony-stimulating factor (G-CSF), comprising four medications. This project initiates a prospective and exploratory clinical study on the DCMG chemotherapy regimen for the treatment of relapsed/refractory AML (Acute Myeloid Leukemia). The study aims to evaluate the efficacy and safety of the DCMG combination chemotherapy regimen in treating relapsed/refractory AML.

ELIGIBILITY:
Inclusion Criteria:

* The patient has fully understood the study, voluntarily agrees to participate, and has signed the Informed Consent Form (ICF);
* Age between 18 and 75 years, with no gender restrictions;
* Confirmed diagnosis of relapsed/refractory AML (Acute Myeloid Leukemia) by pathology (meeting any one of the following criteria):

  1. Patients who meet the diagnostic criteria for acute myeloid leukemia (AML) with minimal residual disease (MRD) positivity;
  2. Or patients who meet the diagnostic criteria for recurrent AML, or refractory AML;
* Serum total bilirubin ≤ 1.5 times the upper limit of normal, serum ALT and AST both ≤ 2.5 times the upper limit of the normal range, serum creatinine ≤ 1.5 times the upper limit of normal;
* Echocardiogram showing left ventricular ejection fraction (LVEF) ≥ 50%;
* Estimated survival time ≥ 3 months;
* ECOG performance status score of 0-2.

Exclusion Criteria:

* The subject's prior anti-tumor treatment history meets one of the following conditions:

  1. Previously received mitoxantrone or mitoxantrone hydrochloride liposome injection;
  2. Previously received doxorubicin or other anthracyclines, with a total cumulative dose of doxorubicin > 360 mg/m² (other anthracycline drugs are converted at a ratio of 1 mg doxorubicin equivalent to 2 mg daunorubicin or 0.5 mg idarubicin);
* Cardiac function and disease meet any of the following conditions:

  1. Long QTc syndrome or QTc interval > 480 ms;
  2. Complete left bundle branch block, second-degree or third-degree atrioventricular block;
  3. Severe, uncontrolled arrhythmia requiring medication;
  4. New York Heart Association (NYHA) classification ≥ Class II;
  5. Ejection fraction (EF) < 50% or below the lower limit of normal for the study center's laboratory;
  6. History of myocardial infarction, unstable angina, severe unstable ventricular arrhythmias, or any other arrhythmia requiring treatment, clinically significant pericardial disease, or evidence on electrocardiogram of acute ischemia or active conduction system abnormalities within 6 months prior to enrollment.
* Underwent any major surgery, radiotherapy, chemotherapy, biological therapy, immunotherapy, or experimental treatment within 2 weeks before the first administration of the study drug;
* Uncontrolled systemic diseases (such as progressive infections, uncontrolled hypertension, diabetes, etc.);
* Previous or current diagnosis of other malignancies (excluding adequately controlled basal cell carcinoma of the skin that is non-melanoma, breast/cervical carcinoma in situ, or other malignancies that have been adequately controlled without treatment in the past five years);
* Active hepatitis B or C infection during the viremic phase (Hepatitis B testing: if either HBsAg or core antibody is positive, add HBV-DNA testing; viral DNA levels exceeding 1x10^3 copies/mL; Hepatitis C testing: if HCV antibody is positive, add HCV-RNA testing; viral RNA levels exceeding 1x10^3 copies/mL);
* Human Immunodeficiency Virus (HIV) infection (HIV antibody positive);
* Pregnant women, breastfeeding women, patients who refuse to use effective contraception during the study period;
* Significant neurological or psychiatric history;
* Patients deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate | At the end of Cycle 2 (each cycle is 28 days)
  Percentage of subjects with complete remission (CR) and incomplete hematologic recovery (CRi)

SECONDARY OUTCOMES:
Relapse-Free Survival | 24 months
  Time interval from leukemia free state to the first recurrence or death
Overall Survival | 24 months
  Time interval from start of treatment until death or last follow-up
Duration of response | Time interval from morphologic/MRD response to loss of response or death
Adverse events | Start of treatment to 2 weeks after end of treatment
  Number of subjects with each adverse event.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No